CLINICAL TRIAL: NCT03527953
Title: Clinical Evaluation of Different Bulk-fill Restorative Resin Restorations
Brief Title: A 24-month Clinical Evaluation of Different Bulk-fill Restorative Resins in Class II Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, A Ruya Yazici, Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 71146310
Record Dates: First submitted 2018-05-05; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Dental Caries
Keywords: bulk-fill restorative resins, dental caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Masking Description: single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tetric EvoCeram BulkFill resin (Active Comparator): Randomly applied
  Interventions: Other: Tetric EvoCeram Bulkfill
- Surefil SDR Flowable bulk-fill resin (Active Comparator): Randomly applied
  Interventions: Other: Surefil SDR Flowable bulkfill
- everX fiber-reinforced resin (Active Comparator): Randomly applied
  Interventions: Other: everX fiber-reinforced resin

INTERVENTIONS:
Other: Tetric EvoCeram Bulkfill — The preparation will be etched with 37% phosphoric acid. It will be then rinsed with an air-water spray and dried, leaving the dentin slightly moist. An etch-and-rinse adhesive, ExciTE F, will be applied and agitated on the prepared surfaces for at least 10 seconds. The adhesive will be air-thinned and light-cured for 20 seconds with an LED curing unit. The sectional matrix will be placed and fixed with wooden wedges. Then the bulk-fill resin composite, TBF, will be placed in bulk in about 4-mm thickness and then will be cured for 20 seconds.
  Arms: Tetric EvoCeram BulkFill resin
Other: Surefil SDR Flowable bulkfill — The preparation will be etched. A two-step etch-and-rinse adhesive, Prime&Bond NT will be applied to all enamel/dentin surfaces, air-dried for 5 seconds, and will be light cured for 10 seconds. After the sectional matrix will be placed, the flowable bulk-fill resin composite, SureFil SDR™ flow (Dentsply Caulk, Milford, DE, USA), will be placed in a 4-mm bulk increment in the dentinal part cured for 20 seconds and will be followed by a covering layer of the nanohybrid resin composite, Ceram.X Mono that will be cured for 20 seconds.
  Arms: Surefil SDR Flowable bulk-fill resin
Other: everX fiber-reinforced resin — The enamel will be etched with 37% phosphoric acid for 10 seconds, then will be rinsed, and dried with an air/water syringe for at least 5 seconds. Self-etch adhesive, G-aenial Bond (GC Co., Tokyo, Japan), will be applied to all enamel/dentin surfaces and gently air thinned and then will be light cured for 10 seconds. After the matrix will be placed and wedged, mesial or distal walls will be built with 1-2-mm layers of G-aenial Posterior resin composite. The fiber-reinforced composite, everX Posterior, will be placed into the cavity in approximately 4-mm thickness. The last 2 mm of the cavity will be restored using the G-aenial Posterior composite as an overlay layer. Each increment will be light cured for 20 seconds using an LED unit.
  Arms: everX fiber-reinforced resin

SUMMARY:
The aim of this study is to evaluate the clinical performance of three different bulk-fill restorative resin materials; a bulk fill resin composite, a flowable bulk fill resin composite and a fiber-reinforced resin in Class II restorations over a period of 24 months.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the 24-month clinical performance of three different bulk-fill restorative resin materials in Class II restorations. Forty patients with at least three approximal lesions in premolar and molar teeth will be participated in the study. A total of 120 Class II cavities will be restored using Tetric EvoCeram Bulk Fill (n=40), SureFil SDR flow + Ceram X mono (n=40), and everX Posterior + G-aenial Posterior (n=40) with their respective adhesives according to the manufacturers' instructions. All restorations will be placed by one operator. The restorations will be evaluated at baseline and at 6, 12, 18, and 24 months using modified USPHS criteria by one examiner. The restoration groups for each category will be compared using Pearson's chi-square test, while Cochran's Q test will be used to compare the changes across different time points within each restorative material (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Patients who accept to participate and sign the informed consent
* Patients who have at least three similar-sized approximal primary caries lesions in premolar and molar teeth.
* The teeth to be restored had a normal occlusal relationship with natural dentition and had adjacent tooth contact and had a normal response to a vitality test with no periapical pathology

Exclusion Criteria:

* Patients who don't accept to participate and sign the informed consent
* Patients who have a history of adverse reaction to the test materials
* Patients who are pregnant or lactating, have fewer than 20 teeth
* Patients who have poor oral hygiene, have severe or chronic periodontal disease, have heavy bruxism

Ages: 20 Years to 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of different restorative resins in class II cavities on posterior teeth according to the modified USPHS criteria | 2 years
  Long-term clinical success of different restorative resins in class II cavities on posterior teeth

CONTACTS AND LOCATIONS:
Overall Officials: A.Ruya Yazici, DDS, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yazici AR, Antonson SA, Kutuk ZB, Ergin E. Thirty-Six-Month Clinical Comparison of Bulk Fill and Nanofill Composite Restorations. Oper Dent. 2017 Sep/Oct;42(5):478-485. doi: 10.2341/16-220-C. Epub 2017 Jun 5. PMID 28581919
- See also: PubMed — http://www.ncbi.nlm.nih.gov/pubmed/28581919?report=abstract